CLINICAL TRIAL: NCT00918645
Title: Measurement of Ca Kinetics in Humans With Prostate Cancer-induced Bone Disease
Brief Title: Calcium-41 (41Ca) Chloride Aqueous Solution in Diagnosing Patients With Prostate Cancer and Bone Metastasis
Acronym: UCDCC#217
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000628784; R21CA127671 (NIH); P30CA093373 (NIH); UCDCC-217 (Other: University of California Davis Cancer Center)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Calcium-41

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 41 Ca (Experimental)
  Interventions: Drug: 41 Ca

INTERVENTIONS:
Drug: 41 Ca — single oral 1.2 microgram dose of 41Ca; the first two recruited study subjects will also receive an oral dose of stable calcium isotope (46Ca) to compare initial kinetics with prior work.
  Other Names: calcium-41 (41Ca) chloride aqueous solution

SUMMARY:
RATIONALE: Diagnostic procedures, such as radionuclide imaging using calcium-41 (41Ca) chloride aqueous solution, may help predict progressive disease in patients with prostate cancer and bone metastasis.

PURPOSE: This clinical trial is studying how well calcium-41 (41Ca) chloride aqueous solution works in diagnosing patients with prostate cancer and bone metastasis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure the pharmacokinetics of a single oral dose of calcium-41 (41Ca) chloride aqueous solution (^41Ca) over 18 months in patients with hormone-refractory prostate cancer and bone metastasis.
* To correlate the ^41Ca-tracer kinetics with time to disease progression, skeletal-related events, and death.

Secondary

* To correlate modulations in baseline urinary ^41Ca clearance with changes in clinically relevant disease parameters, including isotope bone scan data and PSA.
* To combine bone turnover assessments with ^41Ca and collagen/bone cell biomarkers with clinical imaging techniques, especially isotope bone scans, to provide improved stratification of disease stage.

OUTLINE: Patients receive oral calcium-41 (41Ca) chloride aqueous solution (^41Ca) on day 1. Some patients also receive oral calcium-46 (46Ca) chloride aqueous solution (^46Ca).

Urine and blood specimens are collected periodically for 18 months. Blood samples are assayed for bone collagen residues, bone alkaline phosphatase, and PSA. Urine specimens are assessed for ^41Ca/Ca. Isotope bone scintigraphy is use to measure radioactivity.

After completion of study treatment, patients are followed up periodically for 3 years.

ELIGIBILITY:
Eligibility Criteria

* Histologically or cytologically confirmed prostate cancer with a Gleason score available or interpretable
* Prostate cancer deemed to be hormone refractory or androgen independent within the past 12 months
* Evidence of bony metastasis
* Either be receiving bisphosphonate therapy or have received a bisphosphonate within the last 18 months. Participants who are on not on bisphosphonate therapy nor have received it within the last 18 months should currently be on Denosumab therapy. All other anti-cancer therapies are allowed.
* Age >18 years
* ECOG performance status 0-2 (Karnofsky >50%).
* Life expectancy of 6 months or greater.
* Investigators are encouraged to follow good medical practice to assure that all participants have adequate hematologic, hepatic, and renal function.
* Recent or planned isotope bone scan, within 12 months prior to enrollment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Participants will be excluded who have experienced a severe skeletal related event (SRE)within the past 3 months. For this study, an SRE consists of any of the following: palliative radiotherapy to bone, pathologic fractures, spinal cord compression, hypercalcemia of malignancy, and surgery to bone to treat or prevent a fracture.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, chronic kidney disease, hyperthyroidism, or psychiatric illness/social situations that would limit compliance with study requirements.
* Corrected serum calcium <8.0 mg/dL (2.0 mmol/L) or ≥12.0 mg/dL (3.0 mmol/L)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Hillegonds, PhD, Principal Investigator — Lawrence Livermore National Laboratory at University of California; Primo N. Lara, MD, Principal Investigator — University of California, Davis
Locations (1):
- Lawrence Livermore National Laboratory, Livermore, California, United States

REFERENCES:
- See also: Abstract — http://ascopubs.org/doi/abs/10.1200/jco.2012.30.5_suppl.130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 41 Ca
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 41 Ca
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 13
Age, Continuous [Mean (Full Range); unit: Years] | 73.2 [65.0 to 86.1]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Whose Samples Were Measured for Pharmacokinetics
Description: Pre-dose specimens will be provided immediately prior to dose administration. Day 1 specimens shall be collected by the subjects 6 hours after dosing (at home); all subsequent urine specimens may be collected at any time during the day and blood specimens should be taken at the same time of day, if feasible (e.g., morning fasted).
Time Frame: Samples will be collected over 18 months
Population: No data was collected from the specimens.
Arm/Group | 41 Ca
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Patients With Urinary 41Ca Clearance Correlated to Disease Progression
Description: Urinary 41Ca clearance will be measured and correlated with progression by RECIST 1.0 and/or PSA progression of 100% over patient nadir.
Time Frame: Samples will be collected over 18 months
Population: Due to small population size of both Urinary samples and disease progression, no correlation data was collected
Arm/Group | 41 Ca
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With Correlation Between 41Ca Clearance and Disease Stage
Description: Measure baseline 41Ca clearance and correlate with number of baseline bone metastasis lesions.
Time Frame: Samples will be collected over 18 months
Population: Due to small population size Data were not collected
Arm/Group | 41 Ca
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Not required
Description: Patients were followed by good clinical practice guidelines, but toxicities were not recorded for data collection purposes.
Arm/Group | 41 Ca
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This trial was IRB closed after accruing only 13 patients of a potential 30 due to contract period expiring. This termination prior to accrual goal achievement led to small numbers of subjects analyzed with no statistical analysis done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No